CLINICAL TRIAL: NCT03598348
Title: Maintenance Treatment With Capecitabine Plus Apatinib vs. Apatinib and Observation After First-line XELOX/SOX Chemotherapy for Patients With Advanced Gastric Cancer: a Multicenter, Randomized, Controlled Trial
Brief Title: Evaluate the Efficacy of Maintenance Treatment With Capecitabine Plus Apatinib in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianglin Yuan, Professor, Chief physician, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJCC006
Record Dates: First submitted 2017-12-24; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Gastric Cancer
Keywords: advanced gastric cancer, apatinib, capecitabine, maintenance
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Maintenance Treatment Group A (Experimental): Maintenance Treatment with Capecitabine plus Apatinib after First-line XELOX chemotherapy for Patients with Advanced Gastric Cancer
  Interventions: Drug: Apatinib+Capecitabine
- Observation Group (No Intervention): Observation after First-line XELOX chemotherapy for Patients with Advanced Gastric Cancer
- Maintenance Treatment Group B (Experimental): Maintenance Treatment with Apatinib after First-line XELOX chemotherapy for Patients with Advanced Gastric Cancer
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib+Capecitabine — Capecitabine 1000mg/m2 po bid, d1-14, Apatinib 250mg po Qd, Q21d
  Other Names: apatinib; capecitabine
  Arms: Maintenance Treatment Group A
Drug: Apatinib — Apatinib 250mg po Qd
  Arms: Maintenance Treatment Group B

SUMMARY:
This is a multicenter, randomized, controlled trial to evaluate the efficacy and safety of Maintenance Treatment with Capecitabine plus Apatinib, Apatinib and Observation after First-line XELOX/SOX chemotherapy for Patients with Advanced Gastric Cancer

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-75；
2. had histologically confirmed unresectable and/or metastatic (primary or recurrent) adenocarcinoma of the stomach or gastroesophageal junction；
3. received 4-6 cycles of Xelox/SOX regimens as first-line chemotherapy and the response was not progression disease (PD);
4. ECOG 0-2；
5. Patients were tested for tumor HER2 status before treatment, and patients with HER2-negative disease；
6. presence of at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 guidelines；
7. Subjects has to voluntarily join the study and sign the Informed Consent Form for the study;
8. Adequate organ function as defined below: Hematologic ANC ≥ 2*109/L, Platelets ≥ 100*109/L, AST and ALT ≤ 2.5×ULN, TBIL ≤ 1.5×ULN
9. Receiving no form of chemotherapy, targeted therapy or other study medication;

Exclusion Criteria:

1. previous radiotherapy to the abdomen；
2. previous treatment for advanced disease (neoadjuvant chemotherapy was permitted if administered >6 months before enrollment)；
3. pregnant or lactating women or women of childbearing potential；
4. disease progression during the first-line chemotherapy;
5. active gastrointestinal bleeding, arterial thrombosis or cerebrovascular accident within 6 months before enrollment
6. previous treatment of apatinib and Ramucirumab

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2018-01-16 (Actual); Primary Completion 2020-01-16 (Estimated); Study Completion 2020-10-16 (Estimated)

PRIMARY OUTCOMES:
PFS | 36 months
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months

SECONDARY OUTCOMES:
OS | 36 months
  From date of randomization until the date of first documented death from any cause, assessed up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Xianglin Yuan, PhD,MD, Study Chair — Tongji Hospital
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided